CLINICAL TRIAL: NCT05619653
Title: Randomised Placebo Controlled Clinical Trial of Efficacy of MYOcardial Protection in Patients With Postacute inFLAMmatory Cardiac involvEment Due to COVID-19
Brief Title: Myocardial Protection in Patients With Post-acute Inflammatory Cardiac Involvement Due to COVID-19
Acronym: MYOFLAME-19
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Valentina Puentmann (Other)
Collaborators: Bayer (Industry); Alcedis GmbH (Industry)
Responsible Party: Sponsor-Investigator, Valentina Puentmann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYOFLAME-19; 2022-001682-12 (EudraCT Number)
Record Dates: First submitted 2022-11-14; First posted 2022-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Associated Cardiac Involvement; Remodeling, Left Ventricle; Remodeling, Vascular; Left Ventricular Dysfunction; Exercise Intolerance; Vascular Inflammation; Microvascular Angina; Long COVID; Myocarditis, Pericarditis
Keywords: long COVID; postCOVID; endothelial dysfunction; myocarditis
MeSH Terms: conditions — Ventricular Remodeling; Vascular Remodeling; Ventricular Dysfunction, Left; Microvascular Angina; Post-Acute COVID-19 Syndrome; Myocarditis; Pericarditis | interventions — Prednisolone; Losartan

STUDY DESIGN:
Intervention Model Description: multicentre randomised double-blind, placebo-controlled clinical trial 1:1 randomisation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator): Prednisolone and Losartan
  Interventions: Drug: Prednisolone; Drug: Losartan
- Placebo (Placebo Comparator): Placebo 1 and Placebo 2
  Interventions: Drug: Prednisolone; Drug: Losartan

INTERVENTIONS:
Drug: Prednisolone — randomised double-blind, placebo-controlled clinical trial 1:1 randomisation
Drug: Losartan — randomised double-blind, placebo-controlled clinical trial 1:1 randomisation

SUMMARY:
Long COVID or Postacute sequelae of COVID-19 infection (PASC) are increasingly recognised complications, defined by lingering symptoms, not present prior to the infection, typically persisting for more than 4 weeks. Cardiac symptoms due to post-acute inflammatory cardiac involvement affect a broad segment of people, who were previously well and may have had only mild acute illness (PASC-cardiovascular syndrome, PASC-CVS). Symptoms may be contiguous with the acute illness, however, more commonly they occur after a delay. Symptoms related to the cardiovascular system include exertional dyspnoea, exercise intolerance chest tightness, pulling or burning chest pain, and palpitations (POTS, exertional tachycardia).

Pathophysiologically, Long COVID relates to small vessel disease (endothelial dysfunction) vascular dysfunction and consequent tissue organ hypoperfusion due to ongoing immune dysregulation. Active organs with high oxygen dependency are most affected (heart, brain, kidneys, muscles, etc.). Thus, cardiac symptoms are often accompanied by manifestations of other organ systems, including fatigue, brain fog, kidney problems, myalgias, skin and joint manifestations, etc, now commonly referred to as the Long COVID or PASC syndrome.

Phenotypically, PostCOVID Heart involvement is characterised by chronic perivascular and myopericardial inflammation. We and others have shown changes using sensitive cardiac MRI imaging that relate to cardiac symptoms (Puntmann et al, Nature Medicine 2022; Puntmann et al, JAMA Cardiol 2020; Summary of studies included in 2022 ACC PostCOVID Expert Consensus Taskforce Development Statement, JACC 2022, references below).

Early intervention with immunosuppression and antiremodelling therapy may reduce symptoms and development of myocardial impairment, by minimising the disease activity and inducing disease remission. Low-dose maintenance therapy may help to maintain the disease activity at the lowest possible level. The benefits of early initiations of antiremodelling therapy to reduce symptoms of exercise intolerance are well recognised, but not commonly employed outside the classical cardiology contexts, such as heart failure or hypertension. As most patients with inflammatory heart disease only have mild or no structural abnormalities, they are left untreated (standard of care).

The aim of this study is to examine the efficacy of a combined immunosuppressive / antiremodelling therapy in patients with PASC symptoms and inflammatory cardiac involvement determined by CMR, to reduce the symptoms and inflammatory myocardial injury and thereby stop the progression to reduced LVEF, HF and death.

DETAILED DESCRIPTION:
Patients with documented COVID-19 infection, experiencing new cardiac symptoms in the aftermath of COVID-19 infection, fulfilling predefined CMR criteria for PostCOVID myocardial involvement and no previously known or demonstrable cardiovascular disease will be randomised to 16-week treatment with Losartan/Prednisolon or placebo. All imaging is conducted with fidelity to standardised imaging protocol. All images are analysed in a dedicated core-lab to confirm eligibility for inclusion. Investigators and participants remain blinded to group allocation and imaging results.

The primary outcome is a change in LVEF from the baseline to 16 weeks measured by MRI.

Secondary outcomes include changes in clinical symptom scores, imaging parameters, CPET (VO2max), as well as outcomes after 1 years time.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients with documented recent COVID19 infection (>4 weeks)
* PASC Syndrome, defined by persistence or new symptoms, not present prior to the infection.
* CMR evidence of inflammatory cardiac involvement at BL by any of the following criteria:
* Increased native T1≥ 1130 ms at 3.0 Tesla (or 1030 ms at 1.5 Tesla) and/or;
* Increased native T2 ≥39.5 ms at 3.0 Tesla (or 49.5 at 1.5 Tesla) and/or
* present non-ischaemic myopericardial LGE and/or;
* LVEF ≥45 - ≤50%.
* Willingness to comply with the study procedures and study protocol

Exclusion Criteria:

* Severe acute COVID illness requiring hospitalisation
* Known allergy to or intolerance of the study medications
* Symptomatic hypotension (systolic blood pressure less than 90 mm Hg), not reversible with oral hydration
* Any previous or current use of ACE inhibitors, AR Blockers
* Any previous oral prednisolone, or any other immunosuppressive or biological treatment (within prior 10 weeks)
* History or CMR evidence of pre-existing significant heart disease, including:

  1. Known cardiac impairment with LVEF ≤44%
  2. Congestive heart failure (NYHA III-IV)
  3. Active heart failure treatment
  4. Established ischaemic heart disease, peripheral arterial disease and/or cerebrovascular disease
  5. Persistent or permanent atrial fibrillation or significant heart rhythm abnormalities
  6. Congenital or clinically relevant valvular heart disease (moderate or severe)
  7. Specific cardiomyopathy (hypertrophic, hypertensive heart disease, amyloidosis, previous myocarditis, non-ischaemic dilated cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, non-compaction cardiomyopathy, etc).
* Known significant concomitant diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome (e.g. diabetes, lung or hepatic disease, epilepsy, psychiatric disorders, renal disease with a current estimated GFR <30 mL/min/1.73 m² using MDRD formula, chronic systemic infection or immunocompromise)
* Exceeding scanner bore and table-holding capacity: Weight >125 kg, BMI > 35 kg/m2
* Contraindications to contrast-enhanced CMR imaging, e.g.

  1. MR-unsafe implantable device
  2. known allergy to gadolinium-based contrast agent (CBGA)
* For female participants:

  1. Pregnant or breastfeeding women
  2. Persons of childbearing potential not willing to use effective contraception (defined as PEARL index <1 - e.g. contraceptive pill, IUD)
* Known alcohol, drug or chemical abuse
* Patients currently participating in an investigational study or for whom participation is planned.
* Unable to provide written informed consent

Patients with CMR evidence of structural heart disease or incidental heart rhythm abnormalities will be advised to see their own doctor for further investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 16 weeks
  absolute change of LVEF from baseline

SECONDARY OUTCOMES:
Scar burden by late gadolinium enhancement (LGE) | 16 weeks
  mean LGE extent (%) and change thereof from baseline
Cardiopulmonary exercise testing (CPET) | 16 weeks
  Achieved Work rate, VO2max, VCO2 max, RER, AT and Slope and change thereof compared to baseline
Mean T1 and T2 mapping | 16 Weeks
  Mean T1 and T2 mapping values (ms) and absolute change thereof compared to baseline
LV Volume (ml/m2) and LV mass (g/m2) | 16 Weeks
  Average LV Volume (ml/m2) and average LV mass (g/m2) and change there of measures from baseline
LV strain % | 16 Weeks
  absolute change of measures from baseline
Aortic stiffness (PWV) | 16 Weeks
  absolute change of measures from baseline
Aortic wall imaging (LGE) | 16 Weeks
  absolute change of measures from baseline
Average Symptom Score (Modified CCS, NYHA, MRC Dyspnea Score, LC Questionnaire (Sudre et al, NM 2020) | at all available time points compared to baseline
  change thereof compared to baseline
HF and MACE Endpoints | 1 year
  proportion of patients with endpoints
Quality of Life assessment | at all available time points compared to baseline
  Quality of Life assessment (RAND 36-Item health survey V2.0)
Compliance and Tolerance of Therapy | at all available time points compared to baseline
  Compliance and Tolerance of Therapy
Assessment of Treatment Response | 16 weeks
  Number of responders achieving partial or full recovery by imaging markers

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Puntmann, MD, PhD, Principal Investigator — Goethe University Frankfurt; Eike Nagel, MD, PhD, Principal Investigator — Goethe University Frankfurt
Locations (5):
- University Medical Centre Vienna, Vienna, Austria
- Germany (4):
  - Institute for experimental and translational cardiovascular imaging, Frankfurt am Main, Hesse
  - University Hospital Greifswald, Greifswald
  - University Hospital Schleswig-Holstein, Campus KIEL, Kiel
  - University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puntmann VO, Martin S, Shchendrygina A, Hoffmann J, Ka MM, Giokoglu E, Vanchin B, Holm N, Karyou A, Laux GS, Arendt C, De Leuw P, Zacharowski K, Khodamoradi Y, Vehreschild MJGT, Rohde G, Zeiher AM, Vogl TJ, Schwenke C, Nagel E. Long-term cardiac pathology in individuals with mild initial COVID-19 illness. Nat Med. 2022 Oct;28(10):2117-2123. doi: 10.1038/s41591-022-02000-0. Epub 2022 Sep 5. PMID 36064600
- [Background] Writing Committee; Gluckman TJ, Bhave NM, Allen LA, Chung EH, Spatz ES, Ammirati E, Baggish AL, Bozkurt B, Cornwell WK 3rd, Harmon KG, Kim JH, Lala A, Levine BD, Martinez MW, Onuma O, Phelan D, Puntmann VO, Rajpal S, Taub PR, Verma AK. 2022 ACC Expert Consensus Decision Pathway on Cardiovascular Sequelae of COVID-19 in Adults: Myocarditis and Other Myocardial Involvement, Post-Acute Sequelae of SARS-CoV-2 Infection, and Return to Play: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2022 May 3;79(17):1717-1756. doi: 10.1016/j.jacc.2022.02.003. Epub 2022 Mar 16. No abstract available. PMID 35307156
- [Background] Puntmann VO, Carerj ML, Wieters I, Fahim M, Arendt C, Hoffmann J, Shchendrygina A, Escher F, Vasa-Nicotera M, Zeiher AM, Vehreschild M, Nagel E. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Nov 1;5(11):1265-1273. doi: 10.1001/jamacardio.2020.3557. PMID 32730619
- [Background] Puntmann VO, Beitzke D, Kammerlander A, Voges I, Gabbert DD, Doerr M, Chamling B, Bozkurt B, Kaski JC, Spatz E, Herrmann E, Rohde G, DeLeuw P, Taylor L, Windemuth-Kieselbach C, Harz C, Santiuste M, Schoeckel L, Hirayama J, Taylor PC, Berry C, Nagel E. Design and rationale of MYOFLAME-19 randomised controlled trial: MYOcardial protection to reduce post-COVID inFLAMmatory heart disease using cardiovascular magnetic resonance Endpoints. J Cardiovasc Magn Reson. 2025 Summer;27(1):101121. doi: 10.1016/j.jocmr.2024.101121. Epub 2024 Oct 29. PMID 39481808
- See also: Related Info — http://www.cardiac-imaging.org/myoflame-19.html
- See also: Related Info — http://www.myoflame.com/